CLINICAL TRIAL: NCT02507934
Title: 2 Week, Randomized, Double-masked, Controlled, Parallel Group+1 Week Follow-up Study to Evaluate Tolerability, Safety and Efficacy of Lubricin 150 µg/ml vs Sodium Hyaluronate (HA) 0.18% Eye Drops (Vismed®) in Patients With Moderate Dry Eye
Brief Title: Tolerability, Safety and Efficacy of Lubricin Versus Sodium Hyaluronate Eye Drops in Patients With Moderate Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUB0115MD; CIV-15-05-013553 (Other: EudaMed)
Record Dates: First submitted 2015-07-23; First posted 2015-07-24 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The packaging used for the comparator in the present investigation aimed at ensuring a complete masking of the test IMD.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubricin (Experimental): Lubricin 150 μg/ml eye drops solution
  Test investigational device was instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Interventions: Device: Lubricin
- Sodium Hyaluronate (Active Comparator): Vismed®, 0.18% sodium hyaluronate eye drops
  Comparator was instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Interventions: Device: Sodium Hyaluronate

INTERVENTIONS:
Device: Lubricin — Lubricin 150 µg/ml eye drops
  Arms: Lubricin
Device: Sodium Hyaluronate — Sodium hyaluronate 0.18% eye drops
  Other Names: Vismed®
  Arms: Sodium Hyaluronate

SUMMARY:
The objective of this study is to evaluate tolerability, safety and efficacy of Lubricin 150 µg/ml eye drops when compared to a widely used commercial 0.18% sodium hyaluronate eye drop formulation in moderate dry eye patients.

Primary objectives:

* Tolerability using a Visual Analogue Scale (VAS) for foreign body sensation, burning/stinging, itching, pain, stick feeling, blurred vision, and photophobia;
* Treatment-emergent adverse events (TEAEs), assessed throughout the clinical investigation.

Secondary objectives:

* Corneal fluorescein staining (scored using the Oxford scale);
* Schirmer test type I (without anaesthesia);
* Symptom assessment in dry eye (SANDE);
* Ocular protection index (OPI);
* Tear film break-up time (TFBUT);
* Best corrected distance visual acuity (BCDVA);
* Slit lamp examination (SLE) (Eyelid - Meibomian glands, eyelid erythema, eyelid oedema, lashes, conjunctiva erythema, lens, iris, anterior chamber, corneal transparency, corneal neovascularisation);
* Intraocular pressure (IOP);
* Number of instillations of investigational medical device during the second week of the clinical investigation.

All parameters will be evaluated at Screening visit-V1 (Day -7 up to day -5), baseline visit-V2 (Day 1), V3 (Day 7±1), V4 (Day 14±1) and at Final Visit follow-up-V5 (Day 21±1).

DETAILED DESCRIPTION:
This study is a 2 week, randomized, double-masked, controlled, parallel group and 1 week follow-up investigation to evaluate tolerability, safety and efficacy of Lubricin (150 µg/mL) eye drops versus sodium hyaluronate (HA) 0.18% eye drops (Vismed®) in patients with moderate dry eye (DE).

ELIGIBILITY:
Inclusion Criteria:

To be checked at the screening visit (V1) within 7 days before study treatment and confirmed at baseline visit (V2):

1. Patients 18 years of age or older;
2. Patients with moderate dry eye characterized by at least one eye with signs and symptoms of moderate dry eye (grade 2 or 3 of the 2007 DEWS report);
3. Patients diagnosed with dry eye from at least 3 months (current use or recommended use of artificial tears for the treatment of Dry Eye);
4. Average VAS score for typical symptoms of Dry Eye (foreign body sensation, burning/stinging, itching, pain, stick feeling, blurred vision and photophobia) ≥ 25 mm;
5. Corneal staining score with fluorescein > 3 using the Oxford corneal grading system in the worst performing eye;
6. Schirmer test without anaesthesia ≤ 10 mm/5 minutes in the worst performing eye;
7. Tear film break-up time (TBUT) ≤ 10 seconds in the worst performing eye;
8. Best corrected distance visual acuity (BCDVA) score ≥ 0.1 decimal units in both eyes at the time of study enrollment;
9. Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients and/or legal representative must have been approved by the Ethics Committee for the current study.

Exclusion Criteria:

1. Patients with a mild Dry Eye condition (severity level 1 according to the Report of the International Dry Eye Workshop -DEWS, 2007);
2. Patients with a severe Dry Eye condition (severity level 4 according to the Report of the International Dry Eye Workshop -DEWS, 2007);
3. Best corrected distance visual acuity (BCDVA) score of < 0.1 decimal units in either eye at the time of study enrolment;
4. Evidence of an active ocular infection in either eye;
5. History or presence of ocular surface disorders not related to dry eye in either eye;
6. Use of any ocular topical medication other than the study medications for the treatment of ocular diseases including artificial tears during the study period;
7. Use of topical cyclosporine, topical corticosteroids or any other topical medication for the treatment of dry eye in either eye within 30 days of study enrolment;
8. History of any ocular surgery (including laser or refractive surgical procedures) in either eye within the 90 days before study enrolment. Ocular surgery will not be allowed during the study treatment period and elective ocular surgery procedures should not be planned during the duration of the follow-up period;
9. Presence or history of any ocular or systemic disorder or condition that might significantly hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the investigator to be incompatible with the study visit schedule or conduct of trail procedures (e.g. ocular trauma, progressive or degenerative corneal conditions, uveitis, systemic infection.);
10. Known hypersensitivity to one of the components of the study or procedural medications;
11. Participation in another clinical study at the same time as the present study or within 90 days of screening/baseline visit;
12. History of drug, medication or alcohol abuse or addiction;
13. Females of childbearing potential (those who are not surgically sterilized or post-menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

    * are currently pregnant or,
    * have a positive result on the urine pregnancy test at the Screening/Baseline Visit or,
    * intend to become pregnant during the study treatment period or,
    * are breast-feeding or,
    * not willing to use highly effective birth control measures, such as: Hormonal contraceptives - oral, implanted, transdermal, or injected and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or an Intra Uterine Device during the entire course of and 30 days after the study treatment periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2015-10-05 (Actual); Study Completion 2015-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Mantelli, MD-PhD, Study Director — Dompè farmaceutici SpA
Locations (1):
- Dipartimento "Organi di Senso" Università La Sapienza- Policlinico Umberto I, Rome, Italy

REFERENCES:
- [Derived] Lambiase A, Sullivan BD, Schmidt TA, Sullivan DA, Jay GD, Truitt ER 3rd, Bruscolini A, Sacchetti M, Mantelli F. A Two-Week, Randomized, Double-masked Study to Evaluate Safety and Efficacy of Lubricin (150 mug/mL) Eye Drops Versus Sodium Hyaluronate (HA) 0.18% Eye Drops (Vismed(R)) in Patients with Moderate Dry Eye Disease. Ocul Surf. 2017 Jan;15(1):77-87. doi: 10.1016/j.jtos.2016.08.004. Epub 2016 Sep 8. PMID 27614318

RESULTS

PARTICIPANT FLOW:
Groups:
- Lubricin 150 μg/ml: Lubricin 150 μg/ml eye drops solution
  The test investigational device as well as the comparator, was instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Lubricin: Lubricin 150 µg/ml eye drops
- Sodium Hyaluronate 0.18%: Vismed®, 0.18% sodium hyaluronate eye drops
  The comparator, as well as the test investigational device, was instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Sodium Hyaluronate: Sodium hyaluronate 0.18% eye drops
Period: Overall Study
Arm/Group | Lubricin 150 μg/ml | Sodium Hyaluronate 0.18%
Started | 20 | 20
Full Analysis Set Population (FAS) | 19 | 20
Safety Population (SAF) | 20 | 20
Completed | 16 | 20
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) population included all enrolled subjects, who received at least one dose of the IMD (Lubricin or Vismed®) during the treatment phase. This analysis set was used for the efficacy analysis.
Groups:
- Lubricin 150 μg/ml (FAS): Lubricin 150 μg/ml eye drops solution
  The test investigational device as well as the comparator, was instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Lubricin: Lubricin 150 µg/ml eye drops
- Sodium Hyaluronate 0.18% (FAS): Vismed®, 0.18% sodium hyaluronate eye drops
  The comparator, as well as the test investigational device, was instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Sodium Hyaluronate: Sodium hyaluronate 0.18% eye drops
- Total: Total of all reporting groups
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS) | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 28
  >=65 years | 2 | 9 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (11.8) | 61.8 (13.3) | 56.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Foreign Body Sensation, Burning/Stinging, Itching, Pain, Stick Feeling, Blurred Vision, Photophobia and Total Ocular Tolerability Score (VAS)
Description: A global ocular tolerability score was determined using a 100 mm Visual Analogue Scale (VAS) on which 0 meant no symptoms and 100 meant the worst possible discomfort. This evaluation was to be performed before any ophthalmic assessment at each scheduled visit. Specific ocular symptoms were measured with the VAS included: foreign body sensation, burning/stinging, itching, pain, sticky feeling, blurred vision, photophobia. The patients evaluated their symptoms using the VAS giving the value they were feeling from none to an extreme value. The VAS scale was a straight horizontal line of fixed length (100 mm). The ends were defined as the extreme limits of the parameter.
  Please note that Ophthalmological evaluations were performed for both eyes. Hence both the eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: The Full Analysis Set (FAS) population included all enrolled subjects, who received at least one dose of the IMD (Lubricin or Vismed®) during the treatment phase. This analysis set was used for the efficacy analysis. Data in the FAS are analyzed for each eye, left and right respectively. Each eye contributes to the analysis without having defined a study eye.
Measure: Median (Standard Deviation); unit: mm
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
mm
  Foreign body sensation - Left eye - Day 7±1 | -29.3 (27.1) | -16.6 (24.4)
  Foreign body sensation - Right eye - Day 7±1 | -28.4 (29.0) | -20.7 (22.4)
  Foreign body sensation - Left eye - Day 14±1 | -38.9 (23.8) | -23.6 (25.6)
  Foreign body sensation - Right eye - Day 14±1 | -35.9 (23.1) | -24.2 (23.1)
  Foreign body sensation - Left eye - Day 21±1 | -32.7 (29.4) | -23.0 (23.7)
  Foreign body sensation - Right eye - Day 21±1 | -32.3 (26.3) | -23.3 (21.3)
  Burning /Stinging - Left eye - Day 7±1 | -32.1 (30.9) | -23.5 (21.3)
  Burning /Stinging - Right eye - Day 7±1 | -29.2 (28.7) | -27.3 (22.1)
  Burning /Stinging - Left eye - Day 14±1 | -41.9 (26.8) | -31.0 (24.4)
  Burning /Stinging - Right eye - Day 14±1 | -37.9 (27.2) | -33.8 (25.3)
  Burning /Stinging - Left eye - Day 21±1 | -41.2 (27.6) | -29.5 (24.6)
  Burning /Stinging - Right eye - Day 21±1 | -35.7 (25.8) | -32.9 (24.6)
  Itching - Left eye - Day 7±1 | -26.2 (30.6) | -18.2 (22.4)
  Itching - Right eye - Day 7±1 | -18.4 (22.3) | -25.3 (27.2)
  Itching - Left eye - Day 14±1 | -22.5 (21.7) | -31.3 (27.00)
  Itching - Right eye - Day 14±1 | -22.7 (23.2) | -28.5 (26.1)
  Itching - Left eye - Day 21±1 | -21.7 (20.2) | -32.5 (24.6)
  Itching - Right eye - Day 21±1 | -21.9 (23.3) | -29.2 (23.4)
  Pain - Left eye - Day 7±1 | -10.1 (15.2) | -21.0 (29.2)
  Pain - Right eye - Day 7±1 | -7.4 (17.3) | -21.6 (26.4)
  Pain - Left eye - Day 14±1 | -12.4 (15.6) | -22.9 (26.1)
  Pain - Right eye - Day 14±1 | -11.3 (16.6) | -24.9 (27.3)
  Pain - Left eye - Day 21±1 | -12.3 (16.9) | -26.6 (24.0)
  Pain - Right eye - Day 21±1 | -14.3 (15.8) | -25.7 (26.7)
  Sticky feeling - Left eye - Day 7±1 | -28.5 (28.0) | -17.1 (25.3)
  Sticky feeling - Right eye - Day 7±1 | -33.1 (27.8) | -18.0 (21.4)
  Sticky feeling - Left eye - Day 14±1 | -33.1 (30.5) | -21.9 (23.6)
  Sticky feeling - Right eye - Day 14±1 | -35.9 (26.5) | -20.1 (19.3)
  Sticky feeling - Left eye - Day 21±1 | -31.7 (30.8) | -20.2 (26.5)
  Sticky feeling - Right eye - Day 21±1 | -37.3 (26.5) | -19.4 (22.4)
  Blurred vision - Left eye - Day 7±1 | -36.1 (30.4) | -22.7 (21.8)
  Blurred vision - Right eye - Day 7±1 | -28.4 (31.6) | -27.9 (26.2)
  Blurred vision - Left eye - Day 14±1 | -34.9 (25.7) | -27.2 (19.5)
  Blurred vision - Right eye - Day 14±1 | -27.7 (24.9) | -29.0 (22.5)
  Blurred vision - Left eye - Day 21±1 | -37.7 (29.4) | -28.7 (22.6)
  Blurred vision - Right eye - Day 21±1 | -33.3 (26.1) | -33.1 (24.9)
  Photophobia - Left eye - Day 7±1 | -34.9 (33.0) | -26.5 (26.3)
  Photophobia - Right eye - Day 7±1 | -35.2 (29.9) | -28.0 (25.0)
  Photophobia - Left eye - Day 14±1 | -37.0 (30.0) | -29.3 (27.0)
  Photophobia - Right eye - Day 14±1 | -38.6 (27.2) | -30.5 (23.6)
  Photophobia - Left eye - Day 21 ±1 | -42.2 (34.2) | -30.8 (28.0)
  Photophobia - Right eye - Day 21±1 | -39.1 (28.3) | -32.1 (27.6)
  Total - Left eye - Day 7±1 | -189.1 (119.1) | -153.5 (129.1)
  Total - Right eye - Day 7±1 | -179.9 (115.9) | -168.7 (117.3)
  Total - Left eye - Day 14±1 | -220.6 (121.1) | -187.0 (115.3)
  Total - Right eye - Day 14±1 | -209.9 (112.4) | -190.9 (99.7)
  Total - Left eye - Day 21±1 | -219.5 (137.7) | -191.1 (127.4)
  Total - Right eye - Day 21±1 | -213.9 (119.9) | -195.6 (115.9)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Foreign body sensation - Left eye; Test type: Superiority; p = 0.0129, repeated measures ANOVA — For each parameter, for each eye, an ANOVA model for repeated measures has been used by including each available timepoint. The estimated mean difference between treatments (Vismed-Lubricin) over time has been reported and tested; Mean Difference (Final Values) = 8.56, 95% CI 2-sided [2.41 to 14.72]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Foreign body sensation - Right eye; Test type: Superiority; p = 0.0077, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.58, 95% CI 2-sided [1.70 to 13.45]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Burning/ Stinging - Left eye; Test type: Superiority; p = 0.1589, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.99, 95% CI 2-sided [-1.64 to 9.62]
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Burning/ Stinging - Right eye; Test type: Superiority; p = 0.3167, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.78, 95% CI 2-sided [-2.78 to 8.35]
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Itching - Left eye; Test type: Superiority; p = 0.5243, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-7.64 to 3.96]
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Itching - Right eye; Test type: Superiority; p = 0.6714, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [-4.45 to 6.82]
Statistical Analysis 7: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Pain - Left eye; Test type: Superiority; p = 0.0828, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.89, 95% CI 2-sided [-8.31 to 0.53]
Statistical Analysis 8: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Pain - Right eye; Test type: Superiority; p = 0.7823, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-4.77 to 3.62]
Statistical Analysis 9: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Sticky feeling - Left eye; Test type: Superiority; p = 0.0432, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.93, 95% CI 2-sided [0.16 to 9.70]
Statistical Analysis 10: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Sticky feeling - Right eye; Test type: Superiority; p = 0.0088, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.35, 95% CI 2-sided [1.70 to 11.00]
Statistical Analysis 11: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Blurred vision - Left eye; Test type: Superiority; p = 0.0013, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 9.28, 95% CI 2-sided [3.90 to 14.66]
Statistical Analysis 12: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Blurred vision - Right eye; Test type: Superiority; p = 0.00629, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.31, 95% CI 2-sided [-0.30 to 10.92]
Statistical Analysis 13: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Photophobia - Left eye; Test type: Superiority; p = 0.0020, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 9.92, 95% CI 2-sided [3.89 to 15.95]
Statistical Analysis 14: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Photophobia - Right eye; Test type: Superiority; p = 0.0111, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.95, 95% CI 2-sided [1.93 to 13.97]
Statistical Analysis 15: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Total score ocular tolerability - Left eye; Test type: Superiority; p = 0.0448, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 31.67, 95% CI 2-sided [0.78 to 62.56]
Statistical Analysis 16: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Analysis of variance for repeated measures on Total score ocular tolerability - Right eye; Test type: Superiority; p = 0.0834, repeated measures ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 26.36, 95% CI 2-sided [-3.66 to 56.37]

2. Primary Outcome: Treatment-emergent Adverse Events (TEAEs), Assessed Throughout the Study.
Description: TEAEs included all AEs occurring or worsening after the first dose of the IMD. These comprise AEs during the treatment and follow-up period. For TEAE the number of events was provided.
Time Frame: Visit 5/Final visit/Follow up - Day 21±1
Population: The Safety population (SAF)included all subjects who receive at least one dose of the IMDs (Lubricin or Vismed®).
Measure: Number; unit: number of events
Groups:
- Lubricin 150 μg/ml (SAF): Lubricin 150 μg/ml eye drops solution
  The test investigational device as well as the comparator, was instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Lubricin: Lubricin 150 µg/ml eye drops
- Sodium Hyaluronate 0.18% (SAF): Vismed®, 0.18% sodium hyaluronate eye drops
  The comparator, as well as the test investigational device, was instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Sodium Hyaluronate: Sodium hyaluronate 0.18% eye drops
Arm/Group | Lubricin 150 μg/ml (SAF) | Sodium Hyaluronate 0.18% (SAF)
Number analyzed (Participants) | 20 | 20
number of events
  All TEAEs | 3 | 2
  TEAEs - Related to treatment | 0 | 0
  TEAEs - Not related to treatment | 3 | 2
  TEAEs - Mild | 3 | 2
  TEAEs - Moderate | 0 | 0
  TEAEs - Severe | 0 | 0
  Serious TEAEs | 0 | 0
  TEAEs - Leading to discontinuation | 0 | 0

3. Secondary Outcome: Change From Baseline in Corneal Fluorescein Surface Staining (Oxford Score)
Description: The corneal fluorescein staining was graded by using the Oxford scheme to assess cornea and conjunctiva epithelium damage. The Oxford grading scale divides corneal staining into six groups according to severity from 0 (absent) to 5 (severe). The examiner compared the overall appearance of the patient's corneal staining with a reference figure, simulating the pattern of staining encountered in dry eye disease. No attempt was made to count the dots or to assess the position or confluence of the dots. The examiner selected the appropriate grade that best represented the state of corneal staining. The grading system recommended by NEI divides the cornea into five zones (central, superior, temporal, nasal, and inferior) and for each zone, the severity of corneal fluorescein staining is graded on a scale from 0 to 3 based on reference figures. Therefore, the maximum score (worst outcome) was 15, the minimum (best outcome) was 0.
  Please note: both the eyes, right & left, were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
score on a scale
  Left eye - Day 7±1 | -0.8 (0.6) | -0.6 (0.5)
  Right eye - Day 7±1 | -0.7 (0.8) | -0.9 (0.8)
  Left eye - Day 14±1 | -1.4 (1.1) | -0.7 (0.6)
  Right eye - Day 14±1 | -1.5 (0.8) | -0.9 (0.9)
  Left eye - Day 21±1 | -1.8 (1.1) | -0.8 (0.9)
  Right eye - Day 21±1 | -1.8 (0.8) | -1.1 (0.9)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on corneal fluorescein surface staining - Left eye - Day 7 ±1; Test type: Superiority; p = 0.2317, Student t-test for unpaired data; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.14 to 0.57]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on corneal fluorescein surface staining - Right eye - Day 7 ±1; Test type: Superiority; p = 0.6017, Student t-test for unpaired data; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.70 to 0.41]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on corneal fluorescein surface staining - Left eye - Day 14 ±1; Test type: Superiority; p = 0.0232, Student t-test for unpaired data; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [0.11 to 1.36]
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on corneal fluorescein surface staining - Right eye - Day 14 ±1; Test type: Superiority; p = 0.0398, Student t-test for unpaired data; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [0.03 to 1.17]
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on corneal fluorescein surface staining - Left eye - Day 21 ±1; Test type: Superiority; p = 0.0038, Student t-test for unpaired data; Mean Difference (Final Values) = 1.05, 95% CI 2-sided [0.36 to 1.74]
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on corneal fluorescein surface staining - right eye; Test type: Superiority; p = 0.0135, Student t-test for unpaired data; Mean Difference (Final Values) = 0.75, 95% CI 2-sided [0.17 to 1.33]

4. Secondary Outcome: Change From Baseline in Schirmer Test I (Without Anaesthesia)
Description: The Schirmer test type I (without anaesthesia) was performed to measure aqueous tear secretion prior to the instillation of any dilating or anaesthetic eye drops.The rounded bent end of a sterile strip was inserted into the lower conjunctival sac over the temporal one-third of the lower eyelid margin. After 5 minutes had elapsed, the Schirmer"s test strip was removed and the length of the tear absorption on the strip was measured (millimeters/5 minutes). Changes from baseline in values of Schirmer's test type I were summarised by eye and evaluation visit, and stratified by severity level. The longer the wetted length, the healthier the status of the eye.
  Please note that Ophthalmological evaluations were performed for both eyes. Hence both the eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: The Full Analysis Set (FAS) population included all enrolled subjects, who received at least one dose of the IMD (Lubricin or Vismed®) during the treatment phase. Data in the FAS are analyzed for each eye, left and right respectively. Each eye contributes to the analysis without having defined a study eye.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
score on a scale
  Left eye - Day 7±1 | 0.8 (1.3) | 1.4 (2.3)
  Right eye - Day 7±1 | 1.0 (3.0) | 0.8 (2.2)
  Left eye - Day 14±1 | 1.4 (1.4) | 1.4 (2.1)
  Right eye - Day 14±1 | 1.8 (3.9) | 0.5 (2.5)
  Left eye - Day 21±1 | 1.4 (2.2) | 0.3 (3.2)
  Right eye - Day 21±1 | 1.6 (4.1) | 0.4 (2.7)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on Schirmer's test type I strip wetting distance - Left eye - Day 7±1; Test type: Superiority; p = 0.3442, Student t-test for unpaired data; Mean Difference (Final Values) = 0.59, 95% CI 2-sided [-0.66 to 1.83]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on Schirmer's test type I strip wetting distance - Right eye - Day 7±1; Test type: Superiority; p = 0.7720, Student t-test for unpaired data; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-1.99 to 1.49]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on Schirmer's test type I strip wetting distance - Left eye - Day 14±1; Test type: Superiority; p = 0.9725, Student t-test for unpaired data; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-1.49 to 1.44]
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on Schirmer's test type I strip wetting distance - Right eye - Day 14±1; Test type: Superiority; p = 0.2111, Student t-test for unpaired data; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-3.54 to 0.81]
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on Schirmer's test type I strip wetting distance - Left eye - Day 21±1; Test type: Superiority; p = 0.2629, Student t-test for unpaired data; Median Difference (Final Values) = -1.10, 90% CI 2-sided [-3.06 to 0.86]
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline on Schirmer's test type I strip wetting distance - Right eye - 21±1; Test type: Superiority; p = 0.2862, Student t-test for unpaired data; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-3.60 to 1.10]

5. Secondary Outcome: Change From Baseline in SANDE (Symptom Assessment in Dry Eye) - Frequency of Symptoms
Description: The SANDE (Symptom Assessment in Dry Eye) questionnaire was a short questionnaire to evaluate both dry eye frequency and severity by using a 100 mm VAS.
  For the assessment, the subjects marked on the 100 mm VAS line the point that they felt represented their perception of their current state. The VAS score was determined by measuring in millimetres from the left hand end of the line to the point that the subject marked. The SANDE scores was then evaluated for the 2 questions severity (0-100) and frequency (0-100), where 0 was the best condition and 100 marked the worst condition.
  Please note that ophthalmological evaluations were performed for both eyes. Hence both the eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
mm
  Day 7±1 | -29.6 (31.8) | -18.4 (17.8)
  Day 14±1 | -39.6 (29.3) | -21.4 (22.7)
  Day 21±1 | -39.7 (30.9) | -16.2 (22.5)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in symptom assessment in dry eye - Frequency - Day 7±1; Test type: Superiority; p = 0.2075, Student t-test for unpaired data; Mean Difference (Final Values) = 11.24, 95% CI 2-sided [-6.66 to 29.14]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in symptom assessment in dry eye - Frequency - Day 14±1; Test type: Superiority; p = 0.0435, Student t-test for unpaired data; Mean Difference (Final Values) = 18.16, 95% CI 2-sided [0.57 to 35.76]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in symptom assessment in dry eye - Frequency - Day 21±1; Test type: Superiority; p = 0.0133, Student t-test for unpaired data; Mean Difference (Final Values) = 23.58, 95% CI 2-sided [5.24 to 41.93]

6. Secondary Outcome: Change From Baseline in SANDE (Symptom Assessment in Dry Eye) - Severity of Symptoms
Description: The SANDE (Symptom Assessment in Dry Eye) questionnaire was a short questionnaire to evaluate both dry eye severity and frequency by using a 100 mm VAS.
  For the assessment, the subjects marked on the 100 mm VAS line the point that they felt represented their perception of their current state. The VAS score was determined by measuring in millimetres from the left hand end of the line to the point that the subject marked. The SANDE scores were evaluated for the 2 questions severity (0-100) and frequency (0-100), where 0 was the best condition and 100 marked the worst condition.
  Please note that ophthalmological evaluations were performed for both eyes. Hence both the eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
mm
  Day 7±1 | -25.1 (31.2) | -20.7 (2.03)
  Day 14±1 | -37.0 (26.5) | -24.3 (19.2)
  Day 21±1 | -35.8 (29.1) | -22.4 (19.3)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in symptom assessment in dry eye - Severity - Day 7±1; Test type: Superiority; p = 0.6130, Student t-test for unpaired data; Mean Difference (Final Values) = 4.36, 95% CI 2-sided [-12.98 to 21.69]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in symptom assessment in dry eye - Severity - Day 14±1; Test type: Superiority; p = 0.1047, Student t-test for unpaired data; Mean Difference (Final Values) = 12.70, 95% CI 2-sided [-2.78 to 28.18]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in symptom assessment in dry eye - Severity - Day 21±1; Test type: Superiority; p = 0.1108, Student t-test for unpaired data; Mean Difference (Final Values) = 13.40, 95% CI 2-sided [-3.24 to 30.04]

7. Secondary Outcome: Change From Baseline in OPI (Ocular Protection Index)
Description: OPI was used to quantify the interaction between tear film break-up time and blink intervals of a subject. It was based on the idea that, even when the TBUT was normal, if the blink interval was too slow it may cause breakage of tear film due to increased evaporation. The OPI was calculated by dividing TFBUT by inter blink interval (IBI). A visual count of the number of blinks per minute was performed while the subject read the ETDRS chart. ETDRS charts had five Sloan letters on each line; the lines were of equal difficulty, and there was a geometric progression in letter size from line to line. If the IBI and TBUT was same, dividing both give a value of 1.0. If TFBUT was more than IBI, dividing both, gave a value more than 1.0, so dryness would not occur. If TFBUT was less than IBI, dividing both gave a value less than 1.0. A subject was at risk of developing dry eye if the OPI was < 1.0; so the higher the score the better the outcome. Both eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
score on a scale
  Left eye - Day 7±1 | 0.1 (1.0) | 0.3 (0.8)
  Right eye - Day 7±1 | 0.1 (0.8) | 0.4 (0.7)
  Left eye - Day 14±1 | 0.2 (0.9) | 0.0 (0.8)
  Right eye - Day 14±1 | 0.3 (1.1) | 0.0 (0.9)
  Left eye - Day 21±1 | 0.2 (0.8) | -0.2 (0.8)
  Right eye - Day 21±1 | 0.3 (1.1) | -0.1 (0.9)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Ocular Protection Index - Left eye - Day 7±1; Test type: Superiority; p = 0.4980, Student t-test for unpaired data; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.40 to 0.81]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Ocular Protection Index - Right eye - Day 7±1; Test type: Superiority; p = 0.1986, Student t-test for unpaired data; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.18 to 0.83]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Ocular Protection Index - Left eye - Day 14±1; Test type: Superiority; p = 0.4067, Student t-test for unpaired data; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.90 to 0.37]
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Ocular Protection Index - Right eye - Day 14±1; Test type: Superiority; p = 0.5256, Student t-test for unpaired data; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.81 to 0.42]
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Ocular Protection Index - Left eye - Day 21±1; Test type: Superiority; p = 0.1471, Student t-test for unpaired data; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.12 to 0.17]
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Ocular Protection Index - Right eye - Day 21±1; Test type: Superiority; p = 0.2455, Student t-test for unpaired data; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.96 to 0.25]

8. Secondary Outcome: Change From Baseline in TFBUT (Tear Film Break Up Time)
Description: TFBUT was measured by determining the time to tear break-up. The TFBUT test was performed after instillation of 5 µl of 2% preservative-free sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye. With the aid of a slit lamp at 10X magnification using cobalt blue illumination, the examiner monitored the integrity of the tear film, noting the time it took to form lacunae (clear spaces in the tear film) from the time that the eye was opened after the last blink. This measurement was performed within 10 seconds maximum. The TFBUT was measured twice during the first minute after the instillation of the fluorescein. If the 2 readings differed by more than 2 seconds, a third reading was taken. The TFBUT value was the average of the 2 or 3 measurements. Generally, a TFBUT value of 10-35 seconds was considered normal. A value of less than 10 seconds was usually suspicious and may indicate tear film instability. Both the eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
sec
  Left eye - Day 7±1 | 1.8 (2.4) | 1.2 (1.9)
  Right eye - Day 7±1 | 1.2 (2.3) | 1.5 (1.8)
  Left eye - Day 14±1 | 2.7 (2.4) | 0.7 (2.1)
  Right eye - Day 14±1 | 1.9 (2.4) | 0.6 (2.3)
  Left eye - Day 21±1 | 2.6 (2.8) | 0.1 (2.0)
  Right eye - Day 21±1 | 2.1 (2.9) | 0.2 (2.4)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T test p-value - Left eye - Day 7±1; Test type: Superiority; p = 0.4233, Student t-test for unpaired data; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.98 to 0.85]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T test p-value - Right eye - Day 7±1; Test type: Superiority; p = 0.6335, Student t-test for unpaired data; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-1.04 to 1.69]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T test p-value - Left eye - Day 14±1; Test type: Superiority; p = 0.0103, Student t-test for unpaired data; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-3.56 to -0.51]
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T test p-value - Right eye - Day 14±1; Test type: Superiority; p = 0.1006, Student t-test for unpaired data; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.95 to 0.27]
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T test p-value - Left eye - Day 21±1; Test type: Superiority; p = 0.0041, Student t-test for unpaired data; Mean Difference (Final Values) = -2.50, 95% CI 2-sided [-4.15 to -0.85]
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T test p-value - Right eye - Day 21±1; Test type: Superiority; p = 0.0429, Student t-test for unpaired data; Mean Difference (Final Values) = -1.87, 95% CI 2-sided [-3.67 to -0.06]

9. Secondary Outcome: Change From Baseline in BCDVA (Best-corrected Distance Visual Acuity) - ETDRS Score
Description: BCDVA was determined by careful refraction according to the standard protocol for refraction. Chart 1 was used for testing the VA of the right eye; Chart 2 for the left eye; and Chart R for refraction only. Retroilluminated standard Early Treatment of Diabetic Retinopathy Study (ETDRS) charts were used. They had 5 Sloan letters on each line of equal difficulty, and there was a geometric progression in letter size from line to line.VAS awarded one point for every letter correctly guessed. A distance of 4 meters (m) was required between the subject's eyes and the VA chart. When a subject cannot read at least 20 letters on the chart at 4 m, the subject was tested at 1 m. If 20 or more letters were read at 4 m, the VAS for that eye was recorded as the no of letters correct at 4 m plus 30. Otherwise, the VAS was the no of letters read correctly at 1 m plus the no read at 4 m. The higher the score the better the outcome. Both eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
score on a scale
  Left eye - Day 7±1 | 0.2 (0.9) | -0.1 (0.3)
  Right eye - Day 7±1 | 0.3 (0.6) | 0.1 (0.6)
  Left eye - Day 14±1 | -1.7 (7.8) | -0.1 (0.8)
  Right eye - Day 14±1 | -1.0 (8.0) | 0.2 (1.0)
  Left eye - Day 21±1 | 1.1 (1.8) | -0.1 (1.2)
  Right eye - Day 21±1 | 0.9 (2.2) | 0.0 (1.1)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Visual acuity score - Left eye - Day 7±1; Test type: Superiority; p = 0.2338, Student t-test for unpaired data; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.75 to 0.19]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Visual acuity score - Right eye - Day 7±1; Test type: Superiority; p = 0.3081, Student t-test for unpaired data; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.58 to 0.19]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Visual acuity score - Left eye - Day 14±1; Test type: Superiority; p = 0.4287, Student t-test for unpaired data; Mean Difference (Final Values) = 1.59, 95% CI 2-sided [-2.57 to 5.74]
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Visual acuity score - Right eye - Day 14±1; Test type: Superiority; p = 0.5765, Student t-test for unpaired data; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-3.14 to 5.44]
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Visual acuity score - Left eye - Day 21±1; Test type: Superiority; p = 0.0259, Student t-test for unpaired data; Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-2.18 to -0.15]
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Visual acuity score - Right eye - Day 21±1; Test type: Superiority; p = 0.1496, Student t-test for unpaired data; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-2.23 to 0.37]

10. Secondary Outcome: Change From Baseline in Slit Lamp Examination (SLE)
Description: The Slit Lamp Examination was used to examine the structures of the eye (eyelids, lashes, conjunctiva, cornea, lens, iris and anterior chamber) according to different scales: Eyelid - Meibomian glands (from 0-none to 3-severe), Eyelid - Erythema (from 0-none to 4-very severe), Eyelid - Oedema (from 0-none to 4-very severe), Lashes (0-normal 1-abnormal), Conjunctiva - Erythema (from 0-none to 3-severe), Conjunctiva - Oedema (from 0-none to 4-very severe), Lens (from 0-no opacification to 3-severe lens opacification), Iris (0-normal 1-abnormal), Anterior chamber inflammation (from 0-none to 3-severe), Cornea transparency (from 0-completely transparent to 4-complete cornea opacity), Cornea neovascularization (0-absence of neovascularization to 4-neovascularization between 270° and 360°). The higher the score the worse the outcome. There was not a total score.
  Please note: ophthalmological evaluations were performed for both eyes. Hence both eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
score on a scale
  Eyelid - Meibomian glands (Left eye) - Day 7±1 | -0.1 (0.3) | -0.1 (0.3)
  Eyelid - Meibomian glands (Right eye) - Day 7±1 | -0.2 (0.4) | -0.1 (0.2)
  Eyelid - Erythema (Left eye) - Day 7±1 | -0.4 (0.5) | -0.2 (0.4)
  Eyelid - Erythema (Right eye) - Day 7±1 | -0.3 (0.5) | -0.1 (0.2)
  Eyelid - Oedema (Left eye) - Day 7±1 | 0.0 (0.0) | -0.1 (0.2)
  Eyelid - Oedema (Right eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Lashes (Left eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Lashes (Right eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - Erythema (Left eye) - Day 7±1 | -0.4 (0.7) | -0.2 (0.4)
  Conjunctiva - Erythema (Right eye) - Day 7±1 | -0.4 (0.6) | -0.3 (0.4)
  Conjunctiva - Oedema (Left eye) -Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - Oedema (Right eye) -Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Lens (Right eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Lens (Left eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Iris (Left eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Iris (Right eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Left eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Right eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Left eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Right eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Left eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Right eye) - Day 7±1 | 0.0 (0.0) | 0.0 (0.0)
  Eyelid - Meibomian glands (Left eye) - Day14±1 | -0.1 (0.3) | -0.2 (0.4)
  Eyelid - Meibomian glands (Right eye) - Day14±1 | -0.2 (0.4) | -0.1 (0.4)
  Eyelid - Erythema (Left eye) - Day14±1 | -0.6 (0.5) | -0.2 (0.4)
  Eyelid - Erythema (Right eye) - Day14±1 | -0.5 (0.5) | -0.1 (0.3)
  Eyelid - Oedema (Left eye) - Day 14±1 | 0.0 (0.0) | -0.1 (0.2)
  Eyelid - Oedema (Right eye) - Day 14±1 | -0.1 (0.3) | 0.0 (0.0)
  Lashes (Left eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Lashes (Right eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - Erythema (Left eye) - Day 14±1 | -0.9 (0.9) | -0.2 (0.4)
  Conjunctiva - Erythema (Right eye) - Day 14±1 | -0.7 (0.9) | -0.3 (0.4)
  Conjunctiva - Oedema (Left eye) -Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - Oedema (Right eye) -Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Lens (Left eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Lens (Right eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Iris (Left eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Iris (Right eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Left eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Right eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Left eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Right eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Left eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Right eye) - Day 14±1 | 0.0 (0.0) | 0.0 (0.0)
  Eyelid - Meibomian glands (Left eye) - Day 21±1 | -0.2 (0.4) | -0.1 (0.4)
  Eyelid - Meibomian glands (Right eye) - Day 21±1 | -0.2 (0.4) | 0.0 (0.3)
  Eyelid - Erythema (Left eye) - Day 21±1 | -0.8 (0.7) | -0.2 (0.6)
  Eyelid - Erythema (Right eye) - Day 21±1 | -0.6 (0.6) | -0.1 (0.7)
  Eyelid - Oedema (Left eye) - Day 21±1 | -0.1 (0.3) | -0.1 (0.2)
  Eyelid - Oedema ( Right eye) - Day 21±1 | -0.1 (0.3) | 0.0 (0.0)
  Lashes (Left eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Lashes (Right eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - Erythema (Left eye) - Day 21±1 | -0.9 (0.9) | -0.1 (0.6)
  Conjunctiva - Erythema (Right eye) - Day 21±1 | -0.8 (0.7) | -0.2 (0.7)
  Conjunctiva - Oedema (Left eye) -Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Conjunctiva - Oedema (Right eye) -Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Lens (Left eye) - Day 21±1 | -0.1 (0.3) | 0.0 (0.0)
  Lens (Right eye) - Day 21±1 | -0.1 (0.3) | 0.0 (0.0)
  Iris (Left eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Iris (Right eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Left eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Anterior chamber inflammation (Right eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Left eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea transparency (Right eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Left eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
  Cornea neovascularization (Right eye) - Day 21±1 | 0.0 (0.0) | 0.0 (0.0)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Meibomian Glands - Right - Day 7±1; Test type: Superiority; p = 0.2342, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Meibomian Glands - Left - Day 7±1; Test type: Superiority; p = 0.8874, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Erythema - Right - Day 7±1; Test type: Superiority; p = 0.0504, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Erythema - Left - Day 7±1; Test type: Superiority; p = 0.0814, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Oedema - Right - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Oedema - Left - Day 7±1; Test type: Superiority; p = 0.3855, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lashes - Right - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lashes - Left - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Erythema - Right - Day 7±1; Test type: Superiority; p = 0.4754, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Erythema - Left - Day 7±1; Test type: Superiority; p = 0.2914, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Oedema - Right - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Oedema - Left - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lens - Right - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lens - Left - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Iris - Right - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Iris - Left - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Anterior chamber inflammation - Right - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Anterior chamber inflammation - Left - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea transparency - Right - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea transparency - Left - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 21: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea neovascularization - Right - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 22: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea neovascularization - Left - Day 7±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 23: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Meibomian Glands - Right - Day 14±1; Test type: Superiority; p = 0.2429, Wilcoxon (Mann-Whitney)
Statistical Analysis 24: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Meibomian Glands - Left - Day 14±1; Test type: Superiority; p = 0.5707, Wilcoxon (Mann-Whitney)
Statistical Analysis 25: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Erythema - Right - Day 14±1; Test type: Superiority; p = 0.0092, Wilcoxon (Mann-Whitney)
Statistical Analysis 26: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Erythema - Left - Day 14±1; Test type: Superiority; p = 0.0039, Wilcoxon (Mann-Whitney)
Statistical Analysis 27: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Oedema - Right - Day 14±1; Test type: Superiority; p = 0.2882, Wilcoxon (Mann-Whitney)
Statistical Analysis 28: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Oedema - Left - Day 14±1; Test type: Superiority; p = 0.4017, Wilcoxon (Mann-Whitney)
Statistical Analysis 29: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lashes - Right - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 30: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lashes - Left - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 31: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Erythema - Right - Day 14±1; Test type: Superiority; p = 0.0731, Wilcoxon (Mann-Whitney)
Statistical Analysis 32: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Erythema - Left - Day 14±1; Test type: Superiority; p = 0.0020, Wilcoxon (Mann-Whitney)
Statistical Analysis 33: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Oedema - Right - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 34: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Oedema - Left - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 35: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lens - Right - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 36: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lens - Left - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 37: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Iris - Right - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 38: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Iris - Left - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 39: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Anterior chamber inflammation - Right - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 40: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Anterior chamber inflammation - Left - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 41: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea transparency - Right - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 42: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea transparency - Left - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 43: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea neovascularization - Right - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 44: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea neovascularization - Left - Day 14±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 45: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Meibomian Glands - Right - Day 21±1; Test type: Superiority; p = 0.1376, Wilcoxon (Mann-Whitney)
Statistical Analysis 46: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Meibomian Glands - Left - Day 21±1; Test type: Superiority; p = 0.3252, Wilcoxon (Mann-Whitney)
Statistical Analysis 47: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Erythema - Right - Day 21±1; Test type: Superiority; p = 0.0111, Wilcoxon (Mann-Whitney)
Statistical Analysis 48: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Erythema - Right - Day 21±1; Test type: Superiority; p = 0.0049, Wilcoxon (Mann-Whitney)
Statistical Analysis 49: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Oedema - Right - Day 21±1; Test type: Superiority; p = 0.1178, Wilcoxon (Mann-Whitney)
Statistical Analysis 50: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Eyelid - Oedema - Left - Day 21±1; Test type: Superiority; p = 0.9042, Wilcoxon (Mann-Whitney)
Statistical Analysis 51: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lashes - Right - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 52: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lashes - Left - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 53: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Erythema - Right - Day 21±1; Test type: Superiority; p = 0.0253, Wilcoxon (Mann-Whitney)
Statistical Analysis 54: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Erythema - Left - Day 21±1; Test type: Superiority; p = 0.0016, Wilcoxon (Mann-Whitney)
Statistical Analysis 55: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Oedema - Right - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 56: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Conjunctiva - Oedema - Left - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 57: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lens - Right - Day 21±1; Test type: Superiority; p = 0.3165, Wilcoxon (Mann-Whitney)
Statistical Analysis 58: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Lens - Left - Day 21±1; Test type: Superiority; p = 0.3165, Wilcoxon (Mann-Whitney)
Statistical Analysis 59: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Iris - Right - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 60: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Iris - Left - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 61: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Anterior chamber inflammation - Right - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 62: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Anterior chamber inflammation - Left - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 63: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea transparency - Right - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 64: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea transparency - Left - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 65: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea neovascularization - Right - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)
Statistical Analysis 66: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); Wilcoxon Rank Sum Test on changes from baseline in slit lamp examination scores - Cornea neovascularization - Left - Day 21±1; Test type: Superiority; p = 1.0000, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change From Baseline in IOP (Intraocular Pressure)
Description: The intraocular pressure (IOP) of the eye was determined by the balance between the amount of aqueous humor that the eye marked and the ease with which it leaved the eye. IOP was performed using Goldmann applanation tonometry after the instillation of a topical anaesthetic. The Goldmann applanation tonometer measured the force necessary to flatten a corneal area of 3.06 mm diameter. At this diameter, the resistance of the cornea to flattening was counterbalanced by the capillary attraction of the tear film meniscus for the tonometer head. The IOP (in mm Hg) equals the flattening force (in grams) multiplied by 10. IOP was measured in both eyes after completion of all other SLEs to avoid potential interference with the other evaluations. Both eyes were tested. Normal eye pressure was between 10 to 21 mm Hg. High intraocular pressure was greater than 21 mm Hg.
  Please note: ophthalmological evaluations were performed for both eyes. Hence both eyes - right and left - were "study-eyes".
Time Frame: Visit 3 - Day 7±1, Visit 4 - Day 14±1 and Visit 5/Final visit/Follow up - Day 21±1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
mmHg
  Left eye - Day 7±1 | -0.5 (1.6) | 0.7 (1.9)
  Right eye - Day 7±1 | -0.3 (1.8) | 0.2 (1.7)
  Left eye - Day 14±1 | -0.1 (2.5) | 0.2 (2.1)
  RIght eye - Day 14±1 | 0.6 (2.1) | -0.2 (2.0)
  Left eye - Day 21±1 | -0.3 (1.7) | 0.5 (2.0)
  Right eye - Day 21±1 | -0.3 (2.5) | 0.2 (2.6)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Intraocular pressure - Left eye - Day 7±1; Test type: Superiority; p = 0.0599, Student t-test for unpaired data; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [-0.05 to 2.29]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Intraocular pressure - Right eye - Day 7±1; Test type: Superiority; p = 0.3969, Student t-test for unpaired data; Mean Difference (Final Values) = 0.49, 95% CI 2-sided [-0.68 to 1.66]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Intraocular pressure - Left eye - Day 14±1; Test type: Superiority; p = 0.7225, Student t-test for unpaired data; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-1.29 to 1.84]
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Intraocular pressure - Right eye - Day 14±1; Test type: Superiority; p = 0.2690, Student t-test for unpaired data; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-2.14 to 0.62]
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Intraocular pressure - Left eye - Day 21±1; Test type: Superiority; p = 0.2344, Student t-test for unpaired data; Mean Difference (Final Values) = 0.78, 95% CI 2-sided [-0.53 to 2.10]
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on changes from baseline in Intraocular pressure - Right eye; Test type: Superiority; p = 0.5953, Student t-test for unpaired data; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-1.30 to 2.24]

12. Secondary Outcome: Number of Instillations of IMD During the Second Week of the Clinical Investigation
Description: The number of daily instillations of test and comparator IMD from from Visit 3 - Day 7±1 to Visit 4 - Day 14±1
Time Frame: from Visit 3 - Day 7±1 to Visit 4 - Day 14±1
Population: The Full Analysis Set (FAS) population included all enrolled subjects, who received at least one dose of the IMD (Lubricin or Vismed®) during the treatment phase.
Measure: Mean (Standard Error); unit: number of daily administrations
Arm/Group | Lubricin 150 μg/ml (FAS) | Sodium Hyaluronate 0.18% (FAS)
Number analyzed (Participants) | 19 | 20
number of daily administrations
  Day 7: number analyzed (Participants) | 7 | 6
  Day 7 | 4.7 (1.1) | 5.5 (1.0)
  Day 8: number analyzed (Participants) | 17 | 20
  Day 8 | 3.7 (1.5) | 5.1 (1.0)
  Day 9: number analyzed (Participants) | 16 | 20
  Day 9 | 3.9 (1.3) | 4.2 (1.1)
  Day 10: number analyzed (Participants) | 16 | 20
  Day 10 | 3.7 (1.1) | 4.3 (1.0)
  Day 11: number analyzed (Participants) | 16 | 20
  Day 11 | 3.7 (1.0) | 4.4 (1.2)
  Day 12: number analyzed (Participants) | 16 | 20
  Day 12 | 3.4 (1.1) | 4.3 (1.1)
  Day 13: number analyzed (Participants) | 12 | 18
  Day 13 | 3.7 (1.2) | 4.5 (0.9)
  Day 14: number analyzed (Participants) | 9 | 11
  Day 14 | 3.7 (1.3) | 4.2 (1.1)
Statistical Analysis 1: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on number of daily administrations of IMD during the second week of the clinical investigation - Day 7; Test type: Superiority; p = 0.2193, Student t-test for unpaired data; Mean Difference (Final Values) = 0.79, 95% CI 2-sided [-0.54 to 2.11]
Statistical Analysis 2: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on number of daily administrations of IMD during the second week of the clinical investigation - Day 8; Test type: Superiority; p = 0.0024, Student t-test for unpaired data; Mean Difference (Final Values) = 1.34, 95% CI 2-sided [0.51 to 2.18]
Statistical Analysis 3: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on number of daily administrations of IMD during the second week of the clinical investigation - Day 9; Test type: Superiority; p = 0.4250, Student t-test for unpaired data; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.49 to 1.14]
Statistical Analysis 4: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on number of daily administrations of IMD during the second week of the clinical investigation - Day 10; Test type: Superiority; p = 0.1275, Student t-test for unpaired data; Mean Difference (Final Values) = 0.56, 95% CI 2-sided [-0.17 to 1.29]
Statistical Analysis 5: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on number of daily administrations of IMD during the second week of the clinical investigation - Day 11; Test type: Superiority; p = 0.0844, Student t-test for unpaired data; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [-0.09 to 1.42]
Statistical Analysis 6: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on number of daily administrations of IMD during the second week of the clinical investigation - Day 12; Test type: Superiority; p = 0.0238, Student t-test for unpaired data; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [0.12 to 1.60]
Statistical Analysis 7: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on number of daily administrations of IMD during the second week of the clinical investigation - Day 13; Test type: Superiority; p = 0.0369, Student t-test for unpaired data; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.05 to 1.61]
Statistical Analysis 8: Comparison: Lubricin 150 μg/ml (FAS) vs Sodium Hyaluronate 0.18% (FAS); T-test on number of daily administrations of IMD during the second week of the clinical investigation - Day 14; Test type: Superiority; p = 0.3496, Student t-test for unpaired data; Mean Difference (Final Values) = 0.52, 95% CI 2-sided [-0.61 to 1.64]

ADVERSE EVENTS:
Time Frame: The specific period of time over which adverse events data were collected was from day 1 to day 21±1
Description: An Adverse Event (AE) was defined as any untoward medical occurence in a patient or clinical investigation subject administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Groups:
- Lubricin 150 μg/ml (SAF): Lubricin 150 μg/ml eye drops solution
  Both test and comparator were instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Lubricin: Lubricin 150 µg/ml eye drops
- Sodium Hyaluronate 0.18% (SAF): Vismed®, 0.18% sodium hyaluronate eye drops
  Both test and comparator were instilled b.i.d. (two times a day), one drop into each eye, from day 1 to day 7±1 and, then, from 2 to 6 times a day as needed (i.e. prn), one drop into each eye, from day 7±1 to day 14±1.
  After the end of the treatment period, all the subjects used Vismed® 0.18% b.i.d. every 8±1 h, one drop into each eye, from day 14±1 to day 21±1.
  Before the start of the treatment (from day -6/-4 to day -1), the subjects were allowed to use only Nebul®, NaCl 0.9% ocular solution q.i.d. every 4±1 h, one drop into each eye.
  Sodium Hyaluronate: Sodium hyaluronate 0.18% eye drops
Arm/Group | Lubricin 150 μg/ml (SAF) | Sodium Hyaluronate 0.18% (SAF)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubricin 150 μg/ml (SAF) (N=20) | Sodium Hyaluronate 0.18% (SAF) (N=20)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No